CLINICAL TRIAL: NCT06404944
Title: The Use of Implants With a Sloped Platform Edge in Patients With Ridge Atrophy
Brief Title: Using of Implants With a Sloped Platform Edge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI-04
Record Dates: First submitted 2024-04-29; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Bone Resorption
Keywords: Alveolar ridge atrophy; Implant design; Bone loss
MeSH Terms: conditions — Bone Resorption; Bone Diseases, Metabolic | interventions — Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slope Implant (Experimental): The patients received implants with a sloped platform edge.
  Interventions: Procedure: implantation
- Implant and guided bone regeneration (Active Comparator): The patients received implants and guided bone regeneration
  Interventions: Procedure: implantation

INTERVENTIONS:
Procedure: implantation — 1. Incision the mucosa at the alveolar ridge, mucosal-periosteal flap elevation
  2. Placement of the Astra Tech Implant EV Profile (Astra Tech Implant System®; Dentsply Sirona CIS, Sweden)
  3. Placement healing abutment
  4. Suturing the wound tightly
  Arms: Slope Implant
Procedure: implantation — 1. Incision the mucosa at the alveolar ridge, mucosal-periosteal flap elevation
  2. Placement of the Astra Tech OsseoSpeed® TX dental implant (Astra Tech Implant System®; Dentsply Sirona CIS, Sweden)
  3. Guided bone regeneration with xenogeneic bone material Bio-oss® (Geistlich Pharma AG, Sweden) and collagen membrane Bio-Gide® (Geistlich Pharma AG, Sweden)
  4. Suturing the wound tightly
  Arms: Implant and guided bone regeneration

SUMMARY:
An interventional prospective randomized clinical trial (RCT) was conducted in parallel groups. The sample size consisted of 30 patients who were randomly assigned to two groups based on the type of surgical intervention. The first group received implants with a sloped edge platform (Dentsply Sirona CIS, ASTRA TECH Implant System, registered in Russia on 21/12/2019, No. РЗН 2015/3214). The second group received implants with bone grafting. The assessment in the postoperative period included evaluating the condition of the soft tissues, bone resorption, number of analgesics, duration of the operation, edema, keratinized mucosa width, implant stability quotient, pain severity, and quality of life.

DETAILED DESCRIPTION:
The research aimed to compare the clinical and radiological assessment of soft and hard tissues surrounding implants with a sloped edge platform. Thirty patients with alveolar ridge atrophy were examined at the Department of Surgical Dentistry of the E.V. Borovsky Institute of Dentistry, I.M. Sechenov First Moscow State Medical University. These patients displayed a deficiency in hard tissue width, necessitating augmentation for dental implant placement. Patients were randomly divided into two groups based on treatment methods. The first group received implants with a sloped edge platform (Dentsply Sirona CIS, ASTRA TECH Implant System, registered in Russia on 21/12/2019, No. РЗН 2015/3214). The second group underwent treatment with implants of a "standard" design combined with bone grafting. Gender and age characteristics were matched between the groups for comparability.

Patients in the first group were implanted with sloped edge platform implants, while the second group received implants with a different design (Dentsply Sirona CIS, ASTRA TECH Implant System, registered in Russia on 21/12/2019, No. РЗН 2015/3214) incorporating guided bone regeneration. All groups underwent muco-periosteal flap mobilization followed by wound closure without tension using simple interrupted sutures.

In the early postoperative phase, antibacterial and anti-inflammatory therapy was combined with the use of local antiseptics for daily care. Implant uncovering with healing abutment installation occurred 4-6 months post-intervention. The postoperative assessments included evaluating soft tissue condition, bone resorption, analgesic consumption, operation duration, edema, keratinized mucosa width, implant stability quotient, pain severity, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Availability of voluntary informed consent to participate in the study.
2. The presence of an H1I bone defect according to the Cologne classification.
3. Neighboring teeth without hard tissue pathologies and periodontal pathologies.
4. Full sanitation of the oral cavity.

Non-inclusion criteria:

1. The presence of concomitant pathology in the stage of decompensation;
2. Hard smokers (more than 10 cigarettes per day);
3. Radio and chemotherapy in history over the past 5 years;
4. Pregnancy and breastfeeding;
5. Taking medications that affect the healing of soft tissues (nonsteroidal anti-inflammatory drug, steroid drugs).

Exclusion Criteria:

1. Patients with infections either periodontally or periapically, which developed after inclusion in the study;
2. Pregnancy following entrance into the study;
3. Patients having poor oral hygiene or not wanting to carry out oral hygiene measures;
4. Patients who, for one reason or another, could not complete the entire protocol to the end.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
determination of the level of the marginal bone | Day 180 compared to the 0th day (initial value)
  This parameter was determined by analyzing radiovisiography performed on the Vatech EzSensor device (Vatech, South Korea) with an X-ray load of 2μSv 6 months after the operation (after completion of prosthetics). The radiographs were studied using X-ray software on a 27-inch monitor (ASUS) with a screen resolution of 2560 × 1440 pixels. The marginal bone level was assessed using a measuring tool built into the program. The reference point for measurement was the implant shoulder on the medial and distal sides.

SECONDARY OUTCOMES:
Attached mucosa measurement | day 0 (initial value)]
  Evaluation of the width of the keratinized gum will be carried out using a periodontological probe. The width is measured between the mucosal-gingival junction between the vestibular and oral sides.
Attached mucosa measurement | day 180 compared to the 0th day (initial value)
  Evaluation of the width of the keratinized gum will be carried out using a periodontological probe. The width is measured between the mucosal-gingival junction between the vestibular and oral sides.
Evaluation of soft tissue aesthetics | day 180 compared to the 0th day (initial value)]
  Evaluation of soft tissue aesthetics will be carried out according to clinical examination data after the installation of the final orthopedic structure using standard PES (Pink esthetic score). points from 0 to 2, where "2" means a result close to natural.
Assessment of the quality of life | Day 0 (initial value).]
  The patient's quality of life will be assessed using the Oral Health Impact Profile-14 (OHIP-14) questionnaire. points from 0 to 4, where "4" means the worst result
Assessment of the quality of life | Day 1 compared to the 0th day (initial value
  The patient's quality of life will be assessed using the Oral Health Impact Profile-14 (OHIP-14) questionnaire. points from 0 to 4, where "4" means the worst result
Assessment of the quality of life | Day 3 compared to the 0th day (initial value).
  The patient's quality of life will be assessed using the Oral Health Impact Profile-14 (OHIP-14) questionnaire. points from 0 to 4, where "4" means the worst result
Assessment of the quality of life | Day 5 compared to the 0th day (initial value)
  The patient's quality of life will be assessed using the Oral Health Impact Profile-14 (OHIP-14) questionnaire. points from 0 to 4, where "4" means the worst result
Assessment of the quality of life | Day 7 compared to the 0th day (initial value
  The patient's quality of life will be assessed using the Oral Health Impact Profile-14 (OHIP-14) questionnaire. points from 0 to 4, where "4" means the worst result
Assessment of the quality of life | Day 90 compared to the 0th day (initial value)
  The patient's quality of life will be assessed using the Oral Health Impact Profile-14 (OHIP-14) questionnaire. points from 0 to 4, where "4" means the worst result
Assessment of the quality of life | Day 180 compared to the 0th day (initial value
  The patient's quality of life will be assessed using the Oral Health Impact Profile-14 (OHIP-14) questionnaire. points from 0 to 4, where "4" means the worst result
Assessment of consumption of analgesics | Day 1 compared to the 0th day (initial value)
  Patients' analgesic consumption was assessed by estimating the number of packs of Nimesulide (100 mg) taken
Assessment of consumption of analgesics | Day 3 compared to the 0th day (initial value)
  Patients' analgesic consumption was assessed by estimating the number of packs of Nimesulide (100 mg) taken
Assessment of consumption of analgesics | Day 5 compared to the 0th day (initial value)
  Patients' analgesic consumption was assessed by estimating the number of packs of Nimesulide (100 mg) taken
Assessment of consumption of analgesics | Day 7 compared to the 0th day (initial value)
  Patients' analgesic consumption was assessed by estimating the number of packs of Nimesulide (100 mg) taken
Assessment of consumption of analgesics | Day 90 compared to the 0th day (initial value)
  Patients' analgesic consumption was assessed by estimating the number of packs of Nimesulide (100 mg) taken
Assessment of the collateral edema | Day 1 compared to the 0th day (initial value)
  Edema will be clinically assessed by its volume (scores 0-2; 0 points - no edema, 1 point - moderate edema, 2 points - intense edema compared to the condition of adjacent tissues)
Assessment of the collateral edema | Day 3 compared to the 0th day (initial value)
  Edema will be clinically assessed by its volume (scores 0-2; 0 points - no edema, 1 point - moderate edema, 2 points - intense edema compared to the condition of adjacent tissues)
Assessment of the collateral edema | Day 5 compared to the 0th day (initial value)
  Edema will be clinically assessed by its volume (scores 0-2; 0 points - no edema, 1 point - moderate edema, 2 points - intense edema compared to the condition of adjacent tissues)
Assessment of the collateral edema | Day 7 compared to the 0th day (initial value)
  Edema will be clinically assessed by its volume (scores 0-2; 0 points - no edema, 1 point - moderate edema, 2 points - intense edema compared to the condition of adjacent tissues)
Assessment of the severity of pain syndrome | Day 1 compared to the 0th day (initial value)
  Visual Analogue Scale (VAS). Evaluation of the severity of pain syndrome is carried out after surgery using a questionnaire, where : 0 - absence of pain; 1-2 - weak pain; 3-4 - moderate pain; 5-6 - moderate-severe pain; 7-8 - severe pain; 9-10 - unbearable pain.
Assessment of the severity of pain syndrome | Day 3 compared to the 0th day (initial value)
  Visual Analogue Scale (VAS). Evaluation of the severity of pain syndrome is carried out after surgery using a questionnaire, where : 0 - absence of pain; 1-2 - weak pain; 3-4 - moderate pain; 5-6 - moderate-severe pain; 7-8 - severe pain; 9-10 - unbearable pain.
Assessment of the severity of pain syndrome | Day 5 compared to the 0th day (initial value)
  Visual Analogue Scale (VAS). Evaluation of the severity of pain syndrome is carried out after surgery using a questionnaire, where: 0 - absence of pain; 1-2 - weak pain; 3-4 - moderate pain; 5-6 - moderate-severe pain; 7-8 - severe pain; 9-10 - unbearable pain.
Assessment of the severity of pain syndrome | Day 7 compared to the 0th day (initial value)
  Visual Analogue Scale (VAS). Evaluation of the severity of pain syndrome is carried out after surgery using a questionnaire, where: 0 - absence of pain; 1-2 - weak pain; 3-4 - moderate pain; 5-6 - moderate-severe pain; 7-8 - severe pain; 9-10 - unbearable pain
Assessment of the severity of pain syndrome | Day 90 compared to the 0th day (initial value)
  Visual Analogue Scale (VAS). Evaluation of the severity of pain syndrome is carried out after surgery using a questionnaire, where: 0 - absence of pain; 1-2 - weak pain; 3-4 - moderate pain; 5-6 - moderate-severe pain; 7-8 - severe pain; 9-10 - unbearable pain
Operating time estimation | Day 1 compared to the 0th day (initial value)
  The operative time was measured using chronometry from the time of anesthetic administration to the last suture
Implant Stability Quotient (ISQ) | Day 1 compared to the 0th day (initial value)
  The Implant Stability Quotient (ISQ) was measured using Pinguin device (Integration Diagnostics Sweden AB)
Implant Stability Quotient (ISQ) | Day 180 compared to the 0th day (initial value)
  The Implant Stability Quotient(ISQ) was measured using Pinguin device (Integration Diagnostics Sweden AB)

CONTACTS AND LOCATIONS:
Locations (1):
- I.M. Sechenov First Moscow State Medical University (Sechenov University), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
IPD sharing is impossible because of the recommendation of the local ethics committee, the provision of data is possible upon receipt of an official request addressed to the chief researcher